CLINICAL TRIAL: NCT06121024
Title: Long-term Outcomes of Intensive Care Unit Patients With Post-intubation Tracheal Stenosis; 7-year Follow-up
Brief Title: Long-term Outcomes of Post-intubation Tracheal Stenosis; 7-year Follow-up
Status: Completed | Type: Observational
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Collaborators: Yenimahalle Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Onur Kucuk, Department of anesthesiology and reanimation, Principal Investigator, Specialist Doctor, Ankara Ataturk Sanatorium Training and Research Hospital
Other Study IDs: E-2023-52
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Tracheal Stenosis; Intensive Care Unit
Keywords: tracheal stenosis; post-intubation tracheal stenosis; intensive care unit; interventional bronchoscopy
MeSH Terms: conditions — Tracheal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Simple Tracheal Stenosis: Simple stenosis was defined as lesions with a vertical extension <1 cm (short segment) with endoluminal occlusion, without tracheomalacia or loss of cartilage support.
  Interventions: Procedure: Interventional Bronchoscopy
- Complex Tracheal Stenosis: Complex stenosis were defined as lesions ≥1 cm and varying degrees of cartilage involvement or circumferential contractile scar or tracheal stenosis associated with malacia and inflammation.
  Interventions: Procedure: Interventional Bronchoscopy

INTERVENTIONS:
Procedure: Interventional Bronchoscopy — Bronchoscopy offers vital information when evaluating patients suffering from tracheal stenosis. It enables direct visualisation which identifies the lesion, determines its location and extent of airway involvement, highlights vascularity and fragility, allows for tissue diagnosis and enables the operator to assess the extent of mucosal infiltration and airway compression caused by the tumour. The technique facilitates assessment of stenosis diameter for suitable stent selection. In addition to enabling diagnostic bronchoscopy, rigid bronchoscopy offers therapeutic options such as dilatation, cryotherapy and stenting for tracheal stenosis patients. Our clinical setting employs rigid bronchoscopy for interventional procedures with both diagnostic and therapeutic aspects.
  Other Names: Rigid Bronchoscopy

SUMMARY:
This retrospective, observational, cohort study evaluates the treatment management, long-term outcomes and survival analyses in patients hospitalized in the Intensive Care Unit with a diagnosis of Post-Intubation Tracheal Stenosis (PITS) between 1st June 2016 and 1st June 2022. The study emphasizes the role of bronchoscopic interventions in treatment management and the effective and efficient use of health services.

DETAILED DESCRIPTION:
This retrospective study will analyze data from adult patients aged 18 years and above who were admitted with a diagnosis of Post-Intubation Tracheal Stenosis to the intensive care units of Health Sciences University Ankara Atatürk Sanatorium Training and Research Hospital and Yenimahalle Training and Research Hospital between 2016 and 2022. The analysis will examine data from both the hospital registration system and the patients' intensive care files. Patients who have a history of malignancy contributing to tracheal stenosis, patients who have a history of congenital tracheal anomalies or tracheal stenosis, those with incomplete intensive care follow-up information, patient follow-up files or hospital information system data, and patients who have been repeatedly hospitalized (with only the first hospitalisation data taken into account) shall be eliminated from the study. If patients who were discharged from the intensive care unit have one-year post-discharge data, the investigators will obtain the information from the hospital's follow-up system. Otherwise, investigators will collect information by calling patients or patients first-degree relatives by phone.The post-discharge data is from a past period, and the one-year follow-up period for the last patient included in the study ends on 1st June 2023.

The aim of the study is to determine whether early diagnosis and interventional bronchoscopic treatment have an impact on the length of intensive care unit stay and prognosis for patients with Post-Intubation Tracheal Stenosis whilst in the intensive care unit. This will be achieved through an investigation of patient outcomes following appropriate interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18,
* Intensive care patients diagnosed with post-intubation tracheal stenosis (PITS)

Exclusion Criteria:

* Patients with a history of malignancy in the etiology of tracheal stenosis
* Patients with a history of congenital tracheal anomaly or tracheal stenosis
* Patients with missing intensive care follow-up form, patient follow-up file or hospital information system data
* Repeated hospitalizations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective study will analyze data from adult patients aged 18 years and above who were admitted with a diagnosis of PITS to the intensive care units of Health Sciences University Ankara Atatürk Sanatorium Training and Research Hospital and Yenimahalle Training and Research Hospital between 2016 and 2022. Patients who have a history of malignancy contributing to tracheal stenosis, patients who have a history of congenital tracheal anomalies or tracheal stenosis, those with incomplete intensive care follow-up information, patient follow-up files or hospital information system data, and patients who have been repeatedly hospitalized (with only the first hospitalisation data taken into account) shall be eliminated from the study.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2023-11-12 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Mortality | 1 year
  One-year mortality data following interventional bronchoscopic treatment for post-intubation tracheal stenosis in patients hospitalized in the intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Onur KÜÇÜK, specialist, Principal Investigator — Ankara Ataturk Sanatorium Training and Research Hospital
Locations (1):
- Ankara Atatürk Sanatorium Training and Research Hospital, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No